CLINICAL TRIAL: NCT07138586
Title: Evaluation of Low Level Laser Therapy and Lidocaine Versus Chlorhexidine for the Management of Traumatic Oral Ulcers in Children: A Protocol for a Randomized Controlled Study
Brief Title: Evaluation of Low Level Laser Therapy and Lidocaine Versus Chlorhexidine for the Management of Traumatic Oral Ulcers in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0342
Record Dates: First submitted 2025-08-16; First posted 2025-08-24 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-06

CONDITIONS: Traumatic Ulcer of Oral Mucosa
Keywords: traumatic oral ulcer- low level laser therapy- chlorohexidine- lidocaine

STUDY DESIGN:
Intervention Model Description: the study design was a single blinded randomized clinical study
Who Masked: Outcomes Assessor
Masking Description: the outcomes assessor was un aware of the type of treatment given to the patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- low level laser therapy group (Experimental): patients received low level laser therapy using diode laser 980 nm
  Interventions: Radiation: low level laser therapy group
- Lidocaine gel group (Experimental): patients were instructed to use Lidocaine gel (Oracure gel) 4 times daily.
  Interventions: Drug: Lidocaine gel group
- Chlorhexidine mouthwash group (positive control group). (Experimental): patients were instructed to use Chlorhexidine mouthwash (Orovex) 4 times daily (control group).
  Interventions: Drug: Chlorhexidine mouthwash group (positive control group).

INTERVENTIONS:
Radiation: low level laser therapy group — patients received low level laser therapy using diode laser 980 nm with a low power
  Other Names: low level laser therapy- biostimulation
  Arms: low level laser therapy group
Drug: Lidocaine gel group — patients was instructed to use Lidocaine gel (Oracure gel) 4 times daily.
  Other Names: Oracure gel
  Arms: Lidocaine gel group
Drug: Chlorhexidine mouthwash group (positive control group). — patients was instructed to use Chlorhexidine mouthwash (Orovex) 4 times daily (control group).
  Other Names: Orovex mouthwash
  Arms: Chlorhexidine mouthwash group (positive control group).

SUMMARY:
the goal of the study was to evaluate the pain reduction and healing efficiency of traumatic oral ulcers in children using low-level laser therapy with diode laser 980 nm, lidocaine oral gel and chlorhexidine mouthwash

DETAILED DESCRIPTION:
thirty children were randomly allocated to three groups of ten individuals each: Group one: therapy, Group two: using Lidocaine gel 4 times daily and Group three using chlorhexidine mouthwash 4 times daily .

Assessment was done by evaluating pain by Visual Analogue scale; VAS (primary outcome) and assessment of ulcer size by periodontal probe (Secondary outcome) and Parental acceptance of the therapy (tertiary outcome) immediately after treatment, at day two, five, seven, then at two weeks

ELIGIBILITY:
Inclusion Criteria:

* Children from 4-12 years without any apparent medical problem
* Children with history of receiving a dental procedure in the same or the previous day of the onset of ulcer.
* Children having restorations or teeth with sharp edges.
* Children with orthodontic or any other oral appliance.
* No previous treatment with any modality for the ulcer.
* Willingness to participate in the proposed clinical study.

Exclusion Criteria:

* Patients who had psychological or mental diseases.
* Patient under anticoagulants, anti-inflammatory or immunosuppressant medications.
* Children with systemic (endocrine-metabolic) disease; rheumatologic disease; hormone disorder; immunodeficiency; use of corticoid-based therapy.
* Uncooperative children or parents.
* Patients who did not participate twice weekly in the evaluations were excluded

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2025-01-24 (Actual); Primary Completion 2025-04-20 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Subjective pain assessment of the ulcer | 2 weeks
  evaluation of pain associated with the ulcer will be evaluated using visual analoque scale (VAS) before the onset of treatment then follow up of the degree of pain relief associated with treatment

SECONDARY OUTCOMES:
Objective assessment of the ulcer size | 2 weeks
  evaluation of the ulcer size will be done using a graded periodontal probe before the onset of treatment then follow up of the degree of decrease in ulcer size (indicating healing) associated with treatment
Parental satisfaction | 2 weeks
  Parental satisfaction towards treatment procedures, related to duration and frequency of treatment visits will be evaluated using a questionnaire that will be received and answered by the parents at the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maryam m El Mansy, researcher, Principal Investigator — The National Research Centre, Egypt
Locations (1):
- the National research Centre, Dokki, Giza Governorate, Egypt

REFERENCES:
- [Derived] Mansy ME, Rashed MF. Evaluation of low level laser therapy and lidocaine versus chlorohexidine for the management of traumatic oral ulcers in children: a randomized controlled study. Sci Rep. 2026 Jan 27;16(1):3738. doi: 10.1038/s41598-025-34529-8. PMID 41593123